CLINICAL TRIAL: NCT02065102
Title: Optical Coherence Tomography to Improve Clinical Outcomes During Coronary Angioplasty
Status: Completed | Type: Observational
Sponsor: Royal Infirmary of Edinburgh (Other)
Responsible Party: Principal Investigator, Nicholas Cruden, Consultant Cardiologist, Royal Infirmary of Edinburgh
Other Study IDs: 12/R/CAR/13
Record Dates: First submitted 2014-02-12; First posted 2014-02-17 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Angina
Keywords: Rotational atherectomy; Angina; Optical coherence tomography; Intravascular ultrasound; Coronary stent
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Coronary artery stenting has evolved as an effective treatment for angina and involves stretching up narrowings within the heart arteries using a balloon (coronary angioplasty) before implanting a small metal scaffold (stent) to splint the artery open. It is imperative that stents are fully expanded when they are deployed. If not, then patients are exposed to the serious risk of a blood clot forming in the stent (stent thrombosis), or the stent renarrowing (restenosis). One fifth of patients experiencing stent thrombosis will die and 70% will suffer a heart attack. Restenosis is associated with recurrent angina and heart attacks.

Arguably, visualising stents and ensuring adequate stent expansion is most challenging in patients with extensive hardening, or calcification, of the heart arteries. Optical coherence tomography is a novel technique that utilises near-infrared light to look inside small blood vessels in fine detail. It is 10 times more powerful than the best existing technique, intravascular ultrasound.

The purpose of this study is to compare the utility of optical coherence tomography with intravascular ultrasound in patients with heavily calcified heart arteries undergoing rotational atherectomy and coronary stent insertion. It is hoped that the results of this pilot study will provide proof-of-principle and justification for a larger clinical trial to formally assess the role of optical coherence tomography to guide coronary angioplasty and stenting in patients with heavily calcified coronary arteries.

DETAILED DESCRIPTION:
Twelve patients undergoing rotational atherectomy and coronary stenting for angina in Lothian will be recruited. Rotational atherectomy and stent implantation will be performed as part of routine clinical care. Immediately following stent implantation paired intravascular images of the implanted stent will be obtained using both intravascular ultrasound and optical coherence tomography. The stent will then be further dilated at high pressure with a non compliant balloon and the intravascular images repeated with both intravascular ultrasound and optical coherence tomography. The images obtained will be available to the operator to guide further treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing percutaneous coronary intervention requiring rotational atherectomy and coronary stent implantation for calcified coronary artery disease.
* Ability to give informed consent.

Exclusion Criteria:

* Inability to provide informed consent.
* Acute myocardial infarction.
* Cardiogenic shock.
* Renal failure (eGFR <30 mL/min) in patients who are not on dialysis.
* Pregnancy.
* Contrast allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing percutaneous coronary intervention requiring rotational atherectomy and coronary stent implantation in South East Scotland.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Stent malposition expressed as % of total stent area | Day 1
  The amount of stent not in direct contact with the blood vessel wall (malposition) expressed as a % of total stent area.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas L Cruden, MBChB PhD, Principal Investigator — Royal Infirmary of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Lothian, United Kingdom

REFERENCES:
- [Derived] Gudmundsdottir I, Adamson P, Gray C, Spratt JC, Behan MW, Henriksen P, Newby DE, Mills N, Uren NG, Cruden NL. Optical coherence tomography versus intravascular ultrasound to evaluate stent implantation in patients with calcific coronary artery disease. Open Heart. 2015 Dec 22;2(1):e000225. doi: 10.1136/openhrt-2014-000225. eCollection 2015. PMID 26719807